CLINICAL TRIAL: NCT06054867
Title: PRCT002 PRostate Cancer Treatment With the AQUABEAM Robotic System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PROCEPT BioRobotics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CSP0004
Record Dates: First submitted 2023-09-12; First posted 2023-09-26 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Localized Prostate Cancer
Keywords: AQUABEAM; Aquablation; Aquablation therapy; Robotic Waterjet Treatment; RWT; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Aquablation (Experimental)
  Interventions: Device: Robotic Waterjet Treatment

INTERVENTIONS:
Device: Robotic Waterjet Treatment — The Aquablation therapy is a minimally invasive, image-guided, heat-free robotic therapy delivered by the AQUABEAM Robotic System.
  During Aquablation therapy, the AQUABEAM Handpiece is inserted transurethrally into the prostatic urethra. The operating physician then utilizes cystoscopy in conjunction with transrectal ultrasound (TRUS) imaging for real-time visualization. The AQUABEAM Robotic System utilizes high-velocity sterile saline waterjet to resect and remove the prostate tissue according to the operating physician's treatment plan.
  Other Names: Aquablation therapy

SUMMARY:
The goal of this clinical trial is to evaluate the safety of the AQUABEAM Robotic System in treating patients with localized prostate cancer. Participants will go through baseline and follow up assessments up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Stage ≤ T2c
* PSA ≤ 20 ng/ml
* Prostate volume ≥ 30 ml
* Grade Group (GG) 1 or 2: If GG 1: ≥ 3 cores positive for cancer. Note, multiple positive from any MRI targeted lesion will be considered as a single positive core.

Exclusion Criteria:

* Any prior or current treatment for prostate cancer, including but not limited to surgery, radiation therapy (external or brachytherapy), tissue ablation or chemotherapy.
* Patients with previous surgical or minimally invasive treatment of benign prostatic hyperplasia within the prior 12 months.
* Radiographically suspicious lymph node involvement confirmed with biopsy or PET scan.
* Evidence of bone metastasis.
* Evidence of extracapsular involvement.
* Evidence of seminal vesicle invasion on DRE or MRI read as "definite", "probable" or "consistent with"
* Any condition or history of illness or surgery that may pose an additional risk to men undergoing the Aquablation procedure.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who experience a serious device-related adverse event within 12 months following the study treatment. | 12 months post-treatment
  The primary endpoint is the proportion (percentage) of participants who experience a serious device-related adverse event within 12 months following the study treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Southern California, Institute of Urology, Los Angeles, California
  - NorthShore University HealthSystem, Glenview, Illinois
  - NYU Grossman School of Medicine, New York, New York